CLINICAL TRIAL: NCT05403125
Title: Silver Diamine Fluoride: Novel Addition to the Prophylactic Bundle for Dental Management of Radiation-Induced Dental Caries in Oral and Pharyngeal Cancer Patients
Brief Title: SDF Application in Oral Cancer Patients to Prevent Dental Caries
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas A & M University Baylor College Of Dentistry (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Amal Noureldin, Clinical Associate Professor, Texas A & M University Baylor College Of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SDF PCRP
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
Keywords: Oral and Pharyngeal Cancer; Xerostomia; Silver diamine fluoride; Sodium fluoride gel 5000 PPM
MeSH Terms: conditions — Dental Caries; Pharyngeal Neoplasms; Xerostomia

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial, Intention to Treat
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Test and placebo drugs will be identical in appearance and labeled by the manufacturer as A and B. The biostatistician will generate an assignment list. Individual packets will be prepared, and the clinician will open the packet to determine which study drug to apply. The packets and the drug containers will be color coded to minimize error. In each case a second staff member will verify on site that the participant received the correct coded treatment. Blinding: Participants and the examiners will be blind to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Package (Experimental): Topical application of 38% silver diamine fluoride plus 5000 PPM fluoride gel 1 mo before and 1 and 3 months after radiation treatment
  Interventions: Device: silver diamine fluoride, 38%; Device: Sodium fluoride gel, 5000 PPM
- Gel Alone (Active Comparator): Placebo application of silver diamine fluoride plus 5000 PPM fluoride gel 1 mo before and 1 and 3 months after radiation treatment
  Interventions: Device: Sodium fluoride gel, 5000 PPM

INTERVENTIONS:
Device: silver diamine fluoride, 38% — Topical application to all surfaces of the teeth
  Other Names: Advantage Silver Dental Arrest
  Arms: Package
Device: Sodium fluoride gel, 5000 PPM — Gel applied after application of silver diamine fluoride and dispensed for home use
  Other Names: Elevate FluoriMax 5000R

SUMMARY:
The Texas A & M College of Dentistry, with partner Texas Oncology-Baylor Charles A. Sammons Cancer-Center Radiation-Oncology, proposes to conduct a preliminary clinical study (NIH Stage 0) to pilot test a randomized clinical trial of the efficacy of professionally applied 38% silver diamine fluoride to prevent tooth decay in 60 patients who are being treated with radiation for life threatening head and neck cancer.

DETAILED DESCRIPTION:
Head and neck cancer has increased in Texas over the last two decades. Radiation-induced tooth decay is a devastating yet potentially preventable side effect of the cancer treatment. Silver diamine fluoride, already the standard of care in children, is inexpensive, easy to apply, and safe. The objective of the research is to conduct a single site pilot RCT (NIH Stage 0) to determine feasibility and preliminarily assess the efficacy of 38% silver diamine fluoride and 5000 PPM fluoride gel for prevention of radiation-induced dental caries over 6 months. Eligible participants will be up to 60 head and neck cancer patients who are scheduled for radiotherapy. The proposed intervention will be applied within 1 m before and at 1- and 3-m post radiation. The primary outcome is dental caries surfaces at 6 months post-radiotherapy (DMFS).Secondary outcomes are The Gingival Index, Gingival Bleeding Index, MDASI-HN, and Oral Health Quality of Life score will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Head and Neck cancer

Exclusion Criteria:

* Prognosis less than 1 year
* Radiation field of treatment does not involve jaws

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Dental Caries (DMFS) | 6 months
  Dental Caries Surfaces determined by intraoral inspection

SECONDARY OUTCOMES:
Gingival Index | 6 months
  Silness and Loe Gingival Index for assessment of gingival condition (0 to 3) determined clinically
Bleeding Index | 6 months
  Bleeding at 6 sites of each tooth determined clinically
Oral Health Quality of Life | 6 months
  Questionnaire
MD Anderson Symptom Inventory-Head and Neck | 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Amal Noureldin, DDS, Principal Investigator — TAMU Baylor College of Dentistry
Locations (1):
- Baylor College of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No